CLINICAL TRIAL: NCT03712722
Title: Fecal Microbiota Transplantation (FMT) for Recurrent Clostridium Difficile Infection - an Observational Cohort Study
Brief Title: Fecal Microbiota Transplantation (FMT) for Clostridium Difficile
Acronym: CEFTA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Christian Hvas, Associate professor, MD PhD, University of Aarhus
Other Study IDs: 1-16-02-15-16
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Faecal samples, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- rCDI: Adult patients with recurrect Clostridium difficile infection
  Interventions: Other: Faecal microbiota transplantation (FMT)

INTERVENTIONS:
Other: Faecal microbiota transplantation (FMT) — FMT delivered by colonoscopy, nasojejunal tube, glycerol-based capsules, or freeze-dried encapsulated donor faeces

SUMMARY:
Faecal microbiota transplantation (FMT) is used for recurrent Clostridium difficile infection (rCDI) as part of an quality improvement initiative and conducted within the framework of Center for Faecal Microbiota Transplantation at Aarhus University Hospital (CEFTA).

DETAILED DESCRIPTION:
Patients are assessed, treated and monitored at Aarhus University Hospital (AUH) as an Integrated part of the project.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or higher
* documented recurrence of Clostridium difficile

Exclusion Criteria:

* none

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with recurrent Clostridium difficile infection
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Resolution of Clostridium difficile-Associated disease (CDAD) | 8 weeks
  Number of patients with resolution of CDAD, , defined by the absense of diarrhea (3 or fewer bowel movements per day) and formed stools (Bristol 5 or lower) or, in the case of abnormal stool frequency or consistency, a negative Clostridium difficile toxin test week 8

SECONDARY OUTCOMES:
Clinical effect week 8 | 8 weeks
  Number of patients with clinical effect, defined by absense of diarrhea (3 or fewer bowel movements per day) and formed stools (Bristol 5 or lower)
Negative CD test week 8 | 8 weeks
  Number of patients with negative Clostridium difficile toxin test week 8

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No
data access agreement may be made upon request; contact to PI

REFERENCES:
- [Derived] Paaske SE, Baunwall SMD, Rubak T, Ragard N, Kelsen J, Hansen MM, Lodrup AB, Erikstrup LT, Mikkelsen S, Erikstrup C, Dahlerup JF, Hvas CL. Clinical management of Clostridioides difficile infection with faecal microbiota transplantation: a real-world cohort study. EClinicalMedicine. 2025 Jun 19;85:103302. doi: 10.1016/j.eclinm.2025.103302. eCollection 2025 Jul. PMID 40606527
- [Derived] Paaske SE, Baumwall SMD, Rubak T, Birn FH, Ragard N, Kelsen J, Hansen MM, Svenningsen L, Krarup AL, Fernis CMC, Neumann A, Lodrup AB, Glerup H, Vinter-Jensen L, Helms M, Erikstrup LT, Grosen AK, Mikkelsen S, Erikstrup C, Dahlerup JF, Hvas CL. Real-world Effectiveness of Fecal Microbiota Transplantation for First or Second Clostridioides difficile Infection. Clin Gastroenterol Hepatol. 2025 Mar;23(4):602-611.e8. doi: 10.1016/j.cgh.2024.05.038. Epub 2024 Jun 11. PMID 38871148
- [Derived] Baunwall SMD, Hansen MM, Andreasen SE, Eriksen MK, Ragard N, Kelsen J, Grosen AK, Mikkelsen S, Erikstrup C, Dahlerup JF, Hvas CL. Donor, patient age and exposure to antibiotics are associated with the outcome of faecal microbiota transplantation for recurrent Clostridioides difficile infection: A prospective cohort study. Aliment Pharmacol Ther. 2023 Sep;58(5):503-515. doi: 10.1111/apt.17642. Epub 2023 Jul 22. PMID 37482926
- [Derived] Baek OD, Hjermitslev CK, Dyreborg L, Baunwall SMD, Hoyer KL, Ragard N, Hammeken LH, Povlsen JV, Ehlers LH, Hvas CL. Early Economic Assessment of Faecal Microbiota Transplantation for Patients with Urinary Tract Infections Caused by Multidrug-Resistant Organisms. Infect Dis Ther. 2023 May;12(5):1429-1436. doi: 10.1007/s40121-023-00797-y. Epub 2023 Apr 16. PMID 37062804